CLINICAL TRIAL: NCT06967818
Title: Clinical Evaluation of the Combined Effect of a Potassium Nitrate-Based Gel and Diode Laser in the Treatment of Dentin Hypersensitivity: A Randomized Controlled Trial
Brief Title: Combined Use of Potassium Nitrate Gel and Diode Laser for Dentin Hypersensitivity
Acronym: KN-LASER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KNO3LASER
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-08

CONDITIONS: Dentin Hypersensitivity
Keywords: Dentin Hypersensitivity; Potassium Nitrate; Diode Laser; Dental Pain; Desensitizing Treatment; Visual Analog Scale; Schiff Air Index; Laser Therapy; Tooth Sensitivity; Noninvasive Dentistry
MeSH Terms: conditions — Dentin Sensitivity; Toothache | interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium Nitrate Gel + Active Diode Laser (Experimental): Participants receive topical application of a 5% potassium nitrate gel (Emofrom Actisens), followed by treatment with an active 980 nm diode laser (1.5 W/cm² for 1 minute without contact and 1 minute with contact, using a sweeping motion perpendicular to the long axis of the tooth).
  Sensitivity is measured at baseline (T0), immediately after treatment (T1), and at 1 month (T2), 3 months (T3), and 6 months (T4).
  Interventions: Drug: Potassium Nitrate Gel; Device: Diode Laser (Active)
- Potassium Nitrate Gel + Sham Diode Laser (Sham Comparator): Participants receive the same topical application of 5% potassium nitrate gel (Emofrom Actisens), followed by treatment with an inactive (sham) 980 nm diode laser using the same procedure and duration as in the active group, but without laser energy.
  Sensitivity is measured at the same timepoints: baseline (T0), immediately after treatment (T1), 1 month (T2), 3 months (T3), and 6 months (T4).
  Interventions: Drug: Potassium Nitrate Gel; Device: Diode Laser (Sham)

INTERVENTIONS:
Drug: Potassium Nitrate Gel — Topical application of a 5% potassium nitrate gel (Emofrom Actisens) used to treat dentin hypersensitivity.
Device: Diode Laser (Active) — Application of a 980 nm diode laser at 1.5 W/cm² for 1 minute without contact and 1 minute with contact, using a sweeping motion perpendicular to the long axis of the tooth.
  Arms: Potassium Nitrate Gel + Active Diode Laser
Device: Diode Laser (Sham) — Inactive diode laser device used for 1 minute without contact and 1 minute with contact, mimicking the active laser procedure but without energy output.
  Arms: Potassium Nitrate Gel + Sham Diode Laser

SUMMARY:
The aim of this clinical trial is to evaluate the efficacy of the combined use of a diode laser and a potassium nitrate-based desensitizing gel in reducing dentin hypersensitivity in adult patients. Patients who meet the eligibility criteria and for whom informed consent has been obtained will be enrolled and assessed at five timepoints. At baseline (T0), all patients will undergo a professional dental cleaning, collection of medical and dental history, a full periodontal and dental charting, and completion of the Dentine Hypersensitivity Experience Questionnaire (DHEQ) to assess the impact of hypersensitivity on quality of life. Sensitivity will be measured using the Schiff Air Index and the Visual Analog Scale (VAS) in response to air stimulation. At T1, patients will receive the assigned treatment based on randomization. In the test group, the hypersensitive teeth will be treated with topical application of a potassium nitrate gel (Emoform Actisens, 5%) followed by irradiation with a 980 nm diode laser (1.5 W/cm² for 1 minute without contact, then 1 minute with contact and sweeping motion). In the control group, the same potassium nitrate gel will be applied, but the laser will remain inactive (sham laser). Immediately after treatment, the Schiff Air Index and VAS will be reassessed. Follow-up evaluations will be conducted at T2 (1 month after treatment), T3 (3 months), and T4 (6 months). At each follow-up visit, sensitivity will again be measured using the Schiff and VAS indices. At the final follow-up (T4), the DHEQ questionnaire will be administered a second time to assess changes in the patients' perceived impact of dentin hypersensitivity on daily life. Patients are randomized into two groups: Test group: potassium nitrate gel plus active diode laser (980 nm); Control group: potassium nitrate gel plus sham diode laser (inactive). The study aims to determine whether the addition of diode laser irradiation enhances the desensitizing effect of the potassium nitrate gel in both the short and long term (from T1 to T4), as measured by changes in Schiff Air Index, VAS scores, and DHEQ results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good oral hygiene
* Presence of at least one tooth affected by dentin hypersensitivity
* Signed informed consent

Exclusion Criteria:

* Use of analgesic medication
* Ongoing orthodontic treatment
* Non-vital (endodontically treated) teeth
* Teeth with restorative materials on the surface
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Dentin Sensitivity Measured by Schiff Air Index | Baseline (T0), Immediately Post-Treatment (T1), 1 Month (T2), 3 Months (T3), and 6 Months (T4)
  The Schiff Air Index is used to assess sensitivity to evaporative stimuli (air blast). Scores range from 0 to 3, with higher scores indicating greater sensitivity. Measurements will be performed at baseline, immediately after treatment, and during follow-up visits at 1, 3, and 6 months. The primary endpoint is the change in Schiff score from baseline to 6 months.

SECONDARY OUTCOMES:
Change in Pain Perception Measured by Visual Analog Scale (VAS) | Baseline (T0), Immediately Post-Treatment (T1), 1 Month (T2), 3 Months (T3), and 6 Months (T4)
  The VAS is a 10 cm horizontal line on which participants indicate their perceived pain during air stimulus, ranging from 0 (no pain) to 10 (worst imaginable pain). The secondary outcome is the reduction in VAS score between baseline and follow-up visits.
Change in Quality of Life Related to Dentin Hypersensitivity Measured by DHEQ Questionnaire | Baseline (T0) and 6 Months Post-Treatment (T4)
  The Dentine Hypersensitivity Experience Questionnaire (DHEQ) assesses the impact of hypersensitivity on patients' daily lives. It includes 15 items scored from 1 to 7, with a total score range of 15 to 105. Higher scores indicate greater perceived impact. The outcome is the change in total score from baseline to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.